CLINICAL TRIAL: NCT04293913
Title: The Effect of Using Illustrated Communication Material on Anxiety and Comfort in Communication With Patients Receiving Mechanical Ventilator: Randomised Controlled Clinical Trial
Brief Title: Use of Illustrated Material in Communication With the Patient in the Mechanical Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Bircan Kolcak, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16161616
Record Dates: First submitted 2020-02-17; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Comfort; Communication
Keywords: patient; mechanical ventilator; communication material
MeSH Terms: conditions — Anxiety Disorders; Communication

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled clinical trial with two arms: Patients who had undergone cardiac surgery were randomly assigned to intervention (illustrated communication material were used) and control (routine methods in the communication were used) groups when they were connected to the mechanical ventilator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In the intervention group, communication was established with the illustrated communication material. The pain, anxiety scores, and hemodynamic data of the patients were recorded by the intensive care nurse in three consecutive measurements starting with the first communication (0th minute) and at 30th and 60th minutes. On the first postoperative day, the satisfaction of the communication established with them, as well as their evaluations regarding the adequacy of this communication and their comfort levels were determined during the time they received mechanical ventilation therapy.
  Interventions: Behavioral: illustrated communication material
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: illustrated communication material — Illustrated communication material was introduced to the patients in the intervention group. In the process (intensive care) that patients received mechanical ventilation support after the operation, agitation and sedation levels were monitored by the intensive care nurse who was to communicate with the patient using the Richmond Agitation Sedation Scale (RASS). According to this scale, having minimum -2 and maximum +2 points was accepted as the starting criteria for communication (Sessler et al., 2002). Communication was established with the illustrated communication material.
  Arms: intervention group

SUMMARY:
This study was carried out to determine the effect of the use of communication material on the anxiety and comfort of the patient in communication with patients receiving mechanical ventilators.As a result, the use of communication material reduces anxiety and increases patient satisfaction and comfort level. In communicating with intubated patients receiving mechanical ventilator therapy, the use of illustrated communication material is recommended.

DETAILED DESCRIPTION:
The use ofcommunication material in communication with patients receiving mechanical ventilator support increases patient satisfaction and reduces communication difficulties. However, there was no randomized controlled clinical study showing the effect of the use of these materials on patient care outcomes such as anxiety and comfort level.Patients were randomly assigned to the control groups using illustrated communication material and intervention and routine communication methods. The research was carried out in three stages: preoperative, intensive care and one day after surgery. The primary outcomes of the study were pain, anxiety and comfort levels of the patients. Secondary outcomes were the patients' satisfaction with hemodynamic parameters and communication method.

ELIGIBILITY:
Inclusion Criteria:

1. Having undergone cardiac surgery
2. Being applied mechanical ventilator therapy
3. Being 18 or over
4. To have scored minimum 2 to maximum 2 from Richmond Agitation Sedation Scale (RASS)
5. Agree to participate in the research.

Exclusion Criteria:

1. not knowing Turkish
2. Having vision and hearing loss,
3. Having a cognitive or psychological problem that prevents them from communicating. 4. Having an intubation experience before

5. Bleeding, etc. in the early postoperative period. industrial development such as undergoing revision surgery or needing additional sedation,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
change of anxiety over time | The anxiety scores were recorded by the intensive care nurse in three consecutive measurements starting with the first communication (0th minute) and at 30th and 60th minutes
  it was measured by using the Faces Anxiety Scale
comfort level | 1 day after surgery
  Postoperative comfort levels of the patients were determined by the Early Postoperative Comfort Scale.The highest total score that can be obtained from the scale is 144, and the lowest total score is 24. High scores show that comfort is good, and low scores show that comfort is depraved

SECONDARY OUTCOMES:
hemodynamic data | Hemodynamic data were recorded through the patient monitor by intensive care nurses in three consecutive measurements starting with the first communication (0th minute) and at 30th and 60th minutes
  hemodynamic data are systolic and diastolic blood pressure, heart rate, respiration rate, and peripheral oxygen
communication satisfaction and adequacy of communication techniqu, change of pain over time | Pain data were recorded as 30th and 60th minutes, starting from the first communication (0th minute) in mechanical ventilation. Satisfaction and adequacy of communication were evaluated an average of 24 hours after surgery
  It is stated that numerical scales have been adopted more in clinical practice because they are useful in facilitating the definition of pain intensity, facilitating scoring and recording, and evaluating ceiling and floor effects. "The Numerical Evaluation Scale" was used to determine the pain levels of patients and to evaluate their satisfaction with the communication method used and the adequacy of the method

CONTACTS AND LOCATIONS:
Overall Officials: bircan kolcak, lecturer, Principal Investigator — University of Health Sciences, Gulhane Faculty of Nursing, Ankara, Turkey

IPD SHARING:
Plan to Share IPD: Yes
options collected on this subject will be shared in a way that they can be used by other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This work is only available after publication
Access Criteria: it was approved by the responsible researcher of the study to share this study.

REFERENCES:
- [Result] Wang Y, Li H, Zou H, Li Y. Analysis of Complaints from Patients During Mechanical Ventilation After Cardiac Surgery: A Retrospective Study. J Cardiothorac Vasc Anesth. 2015 Aug;29(4):990-4. doi: 10.1053/j.jvca.2015.01.036. Epub 2015 Jan 29. PMID 25939965
- [Derived] Kolcak B, Ayhan H, Tastan S. The effect of using illustrated materials for communication on the anxiety and comfort of cardiac surgery patients receiving mechanical ventilator support: A randomized controlled trial. Heart Lung. 2023 May-Jun;59:157-164. doi: 10.1016/j.hrtlng.2023.02.005. Epub 2023 Feb 22. PMID 36827715

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT04293913/Prot_SAP_ICF_000.pdf